CLINICAL TRIAL: NCT03024580
Title: A Pilot Study Evaluating Megestrol Acetate Modulation in Advanced Breast Cancer With Positive Hormonal Receptor
Brief Title: A Study Evaluating Megestrol Acetate Modulation in Hormone Receptor Positive Advanced Breast Cancer
Acronym: MEGA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Collaborators: Cancer Research UK Cambridge Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 64/16
Record Dates: First submitted 2017-01-04; First posted 2017-01-19 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Breast Neoplasm
Keywords: Megestrol Acetate; Steroid, Receptors
MeSH Terms: conditions — Breast Neoplasms | interventions — Megestrol Acetate; Tablets; Anastrozole; Letrozole; exemestane; Tamoxifen; Fulvestrant; Solutions; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Megestrol acetate (Experimental): Megestrol acetate 160 mg PO daily until disease progression or unacceptable toxicity Tumor biopsy and blood collection before treatment initiation and at the time of disease progression.
  Interventions: Drug: Megestrol Acetate 160Mg Tablet
- Anastrozole (Active Comparator): Anastrozole 1 mg PO daily until disease progression or unacceptable toxicity Tumor biopsy and blood collection before treatment initiation and at the time of disease progression.
  Interventions: Drug: Anastrozole 1Mg Tablet
- Letrozole (Active Comparator): Letrozole 2.5 mg PO daily until disease progression or unacceptable toxicity Tumor biopsy and blood collection before treatment initiation and at the time of disease progression.
  Interventions: Drug: Letrozole 2.5Mg Tablet
- Exemestane (Active Comparator): Exemestane 25 mg PO daily until disease progression or unacceptable toxicity Tumor biopsy and blood collection before treatment initiation and at the time of disease progression.
  Interventions: Drug: Exemestane 25 MG
- Tamoxifen (Active Comparator): Tamoxifen 20 mg PO daily until disease progression or unacceptable toxicity Tumor biopsy and blood collection before treatment initiation and at the time of disease progression.
  Interventions: Drug: Tamoxifen 20Mg Tablet
- Fulvestrant (Active Comparator): Fulvestrant 500 mg intramuscularly (IM) d1, d14, d28 and q28 days until disease progression or unacceptable toxicity Tumor biopsy and blood collection before treatment initiation and at the time of disease progression.
  Interventions: Drug: Fulvestrant 50Mg Solution for Injection

INTERVENTIONS:
Drug: Megestrol Acetate 160Mg Tablet — Megestrol acetate 160 mg PO daily
  Other Names: MA
  Arms: Megestrol acetate
Drug: Anastrozole 1Mg Tablet — Anastrozole 1 mg PO daily OR
  Other Names: Anastrozole
  Arms: Anastrozole
Drug: Letrozole 2.5Mg Tablet — Letrozole 2.5 mg PO daily OR
  Other Names: Letrozole
  Arms: Letrozole
Drug: Exemestane 25 MG — Exemestane 25 mg PO daily
  Other Names: Exemestane
  Arms: Exemestane
Drug: Tamoxifen 20Mg Tablet — Tamoxifen 20 mg PO daily
  Other Names: Tamoxifen
  Arms: Tamoxifen
Drug: Fulvestrant 50Mg Solution for Injection — Fulvestrant 500 mg IM d1, d14, d28 and q28 days
  Other Names: Fulvestrant
  Arms: Fulvestrant

SUMMARY:
This pilot trial evaluates in vivo megestrol acetate (MA) modulation of steroidal receptors in advanced breast cancer.

DETAILED DESCRIPTION:
Progesterone receptor (PR) expression has been considered a biomarker of oestrogen receptor-α (ERα) activity. This longstanding relationship has been recently challenged and instead of being merely an ERα-induced gene target, PR may be a critical determinant of ERα activity. The functional significance of this steroid receptor crosstalk is regulation of a gene expression program associated with low tumorigenicity; hence, better disease outcome. Genomic alterations in the PR genomic locus seem to be a relatively common mechanism for reduction of PR expression, which may consequently lead to altered ERα chromatin binding and target gene expression patterns that increase breast tumorigenicity and confers a poor clinical outcome. This ERα-PR crosstalk may be directly influenced by many variables, including the relative receptor levels and the hormonal milieu.

ER-positive advanced breast cancer is a heterogeneous group of diseases with considerable variability in outcome to a range of treatments. Prior response predicts the likelihood of subsequent benefit from another endocrine agent and this should be taken into account in the treatment decision process when assessing whether to prescribe a subsequent endocrine therapy. Despite the enormous progress made regarding the elucidation of breast cancer subgroups and their molecular drivers, most information comes from primary tumors. MA lacks cross-resistance and is active after acquired resistance to potent AI. This pilot trial evaluates in vivo MA modulation of steroidal receptors in advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic breast cancer with ER and/or PR positive (primary tumor)
* Metastatic site amenable to biopsy

Exclusion Criteria:

* Platelet count below 100,000 / mm3
* Renal or hepatic impairment
* Coagulation disorder

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03-06 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From date of randomization until disease progression or death due to any cause, assessed up to 18 months
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 18 months

SECONDARY OUTCOMES:
Overall survival | From date of randomization until death, assessed up to 18 months
  From date of randomization until the date of death from any cause, assessed up to 18 months
Clinical benefit | Partial response and stable disease for more than 24 weeks, assessed up to 18 months
  Partial response and stable disease for more than 24 weeks, as per RECIST criteria, from date of randomization until the date of first documented progression or date of death, whichever came first, assessed up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: José Bines, MD, PhD, Study Chair — Instituto Nacional de Cancer, Brazil; Jason Carroll, PhD, Study Chair — Cancer Research UK Cambridge Institute
Locations (1):
- Hospital do Cancer III, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No